CLINICAL TRIAL: NCT01025700
Title: A Double-Blind Placebo Control Study on the Use of Nabilone for Outpatient Management of Acute Marijuana Withdrawal
Brief Title: Nabilone & Marijuana Addiction
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Shaohua Lu, MD, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H08-01999
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Marijuana Smoking
Keywords: Efficacy; Marijuana; Reduction; Craving
MeSH Terms: conditions — Marijuana Smoking; Marijuana Abuse | interventions — nabilone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cesemat (Experimental)
  Interventions: Drug: Cesemat
- Placebo (No Intervention)

INTERVENTIONS:
Drug: Cesemat — 1 mg capsule per day for 21 days
  Other Names: Nabilone
  Arms: Cesemat

SUMMARY:
Safety of Nabilone in reducing marijuana craving

DETAILED DESCRIPTION:
Randomized double blind trial into the safety and efficacy of Cesemat for the treatment of marijuana use

ELIGIBILITY:
Inclusion Criteria:

* 19 years or older
* History of marijuana use

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability to Nabilone

SECONDARY OUTCOMES:
Marijuana craving questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Shaohua Lu, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital - Psychiatry Outpatient, Vancouver, British Columbia, Canada